CLINICAL TRIAL: NCT05998616
Title: The Feasibility and Efficacy of a Remotely Delivered Exercise Training Intervention for the Hispanic/Latino Community With Multiple Sclerosis
Brief Title: Feasibility of Remote Exercise Training for Hispanics/Latinos With MS
Acronym: FERLAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Robert W Motl, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Study2023-0665; P50MD017349 (NIH)
Record Dates: First submitted 2023-08-01; First posted 2023-08-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Hispanics/Latinos; Exercise Intervention; Remote Exercise Training; Feasibility Study; Randomized Controlled Trial; Health Disparities; Social Determinants of Health; Physical Function; Cognitive Function; Fatigue; Quality of Life; Telerehabilitation; Health Equity
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Intervention Model Description: FERLA MS is a parallel-group, randomized controlled trial, where eligible participants with MS will be randomly assigned to either the remotely-delivered exercise intervention group or the remotely-delivered and supported flexibility control group. Both groups will receive intervention materials and support via teleconferencing or phone calls. The exercise group will follow a theory-based aerobic and resistance training program, while the control group will engage in flexibility exercises.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and outcomes assessors will be blinded to participant group assignment (exercise intervention or flexibility control group). However, it is important to note that due to the nature of the intervention, participants and outcomes assessors will be aware of the type of intervention received (aerobic/resistance training exercise or flexibility exercises). This is because the exercise intervention and flexibility control involve different activities. Randomization will be conducted by the investigator, who will not be involved in consent, delivery intervention, data collection, and outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training Program (Experimental): Participants will receive a theory-based, remotely-delivered exercise training program that includes aerobic and resistance exercise training.
  Interventions: Behavioral: Exercise Training Program
- Flexibility Program (Active Comparator): Participants will receive a remotely-delivered flexibility program, focusing on improving flexibility and range of motion.
  Interventions: Behavioral: Flexibility Program

INTERVENTIONS:
Behavioral: Exercise Training Program — The intervention group will be encouraged to complete aerobic and resistance training exercises three times a week, and either at home, in the community (e.g., park, shopping mall), or any suitable environment of the participant's choice. Exercise equipment for monitoring walking and complete resistance training will be provided to the intervention group. The exercise training prescription involves 30+ minutes of moderate-intensity walking (≥100 steps/min) monitored by a waist-worn pedometer, and resistance training consisting of 1-2 sets, 10-15 repetitions of 5-10 exercises targeting lower and upper body, and core muscle groups using elastic bands.
  Arms: Exercise Training Program
Behavioral: Flexibility Program — The control group will be encouraged to complete stretching and range of motion exercises three times a week, and either at home, in the community (e.g., park, shopping mall), or any suitable environment of the participant's choice. Exercise equipment (yoga mat) for monitoring walking and complete flexibility training will be provided to the control group. The flexibility training prescription involves stretches from the Stretching for People with MS: An Illustrated Manual from the National MS Society.
  Arms: Flexibility Program

SUMMARY:
The goal of this clinical trial is to investigate the potential benefits of a specially designed exercise program for Hispanics/Latinos with multiple sclerosis (MS). The main questions it aims to answer are:

* Can a 4-month remotely-delivered exercise training program improve physical function, symptom management, and quality of life in Hispanics/Latinos with MS?
* How do social determinants of health, such as income, education, access to healthcare, and social support, influence the feasibility and effectiveness of the exercise intervention?

Participants in this study will engage in a 4-month remotely-delivered exercise training intervention that includes flexibility, or aerobic and resistance exercise training sessions. They will work with experienced coaches who will guide and support them throughout the program. The researchers will compare the participants who receive the exercise intervention with a control group to see if the exercise program leads to significant improvements in physical function, fatigue, mood, and overall well-being for Hispanics/Latinos with MS. The study aims to empower this underserved population and provide insights for future healthcare and research initiatives.

DETAILED DESCRIPTION:
The FERLA MS study is a randomized controlled trial aimed at investigating the feasibility and effectiveness of a remotely-delivered exercise training intervention for Hispanics/Latinos with MS. This study aims also aims to address the significant health disparities faced by this underserved population and provide insights into the potential benefits of exercise training in managing MS symptoms and improving quality of life.

Multiple sclerosis (MS) is an autoimmune disease of the central nervous system, affecting millions of adults in the United States. Hispanics/Latinos with MS are particularly vulnerable to more aggressive disease progression and greater long-term disability compared to other racial/ethnic groups. These disparities are likely influenced by social determinants of health (SDOH), such as limited access to healthcare, medical services, and underrepresentation in medical research. The FERLA MS study seeks to explore the role of exercise training as a disease-modifying and symptom-managing intervention for enhancing health outcomes and overall well-being in this marginalized population.

The study has three main aims:

Aim #1: Assess the Feasibility of the Exercise Intervention. This aim focuses on evaluating the feasibility of a 4-month remotely-delivered exercise training intervention for Hispanics/Latinos with MS. The research team will assess the process, resource, management, and scientific measures to determine the practicality, safety, and efficacy of the intervention.

Aim #2: Evaluate the Efficacy of the Exercise Intervention. The second aim involves evaluating the effectiveness of the exercise intervention in improving physical function, symptom management, and overall quality of life compared to an active control condition. Specific outcomes include the 30-second sit-to-stand test, neuropsychological measures of cognition, fatigue, depression, anxiety, and self-reported health-related quality of life.

Aim #3: Explore the Impact of SDOH Factors. The third aim is to explore the influence of SDOH, such as income, education, access to healthcare, and social support, on the feasibility and potential efficacy of the exercise intervention for improving outcomes in Hispanics/Latinos with MS.

The study is guided by the following hypotheses:

Hypothesis 1: The remotely-delivered exercise training intervention will be feasible for Hispanics/Latinos with MS, as evidenced by high recruitment, enrollment, adherence, and retention rates, along with reasonable time, space, and monetary costs, and safe and effective delivery leading to improvements in MS symptoms and outcomes.

Hypothesis 2: Participants in the intervention condition will demonstrate significant improvements in physical function, cognition, fatigue, mood, and quality of life compared to the active control.

Hypothesis 3: Social determinants of health will significantly influence the feasibility and effectiveness of the exercise intervention in improving physical and mental health outcomes for Hispanics/Latinos with MS.

The FERLA MS study follows a parallel group, randomized controlled trial design. Eligible participants will be randomly assigned to either the remotely-delivered exercise intervention condition or the control condition. The exercise intervention will be based on the Guidelines for Exercise in Multiple Sclerosis (GEMS) and will include both aerobic and resistance training sessions. Aerobic Exercise: Participants will engage in moderate-intensity walking for 30+ minutes three days per week. The progression of the aerobic exercise will follow different trajectories based on individual needs and abilities. Resistance Exercise: The resistance training will consist of 1-2 sets of 10-15 repetitions of 5-10 exercises targeting different muscle groups, performed three days per week using elastic resistance bands. One-on-One Coaching: The exercise program involves one-on-one semi-structured sessions with MS exercise specialists (behavioral coaches) who will provide guidance, oversight, and support to participants. Coaches will also help with action planning, self-monitoring, and deliver content-relevant newsletters based on social cognitive theory. Control Condition: Participants in the control condition will engage in flexibility exercises through telerehabilitation, aimed at improving range of motion and stretching.

The primary endpoint is the feasibility of the remotely-delivered exercise program. Secondary outcomes include physical function, cognitive function, fatigue, mood, and health-related quality of life. The study will also explore the impact of social determinants of health as tertiary outcomes.

Participants' total time commitment for the study will be approximately 5 months, including recruitment, screening, baseline measures, the 4-month exercise or control intervention, and post-intervention measures. Enrollment duration for all study subjects is anticipated to take approximately 2-3 months, with the study projected to be completed by December 1, 2024. Participants must be aged between 18-65 years, diagnosed with MS, relapse-free for at least 30 days, able to walk with or without an assistive device, have no contraindications to exercise, and self-identify as Hispanic/Latino. Individuals with severe cognitive impairments, other neurological conditions, or medical conditions limiting exercise participation will be excluded.

The FERLA MS study will be conducted in compliance with all relevant institutional review board (IRB) regulations and ethical principles outlined in the Declaration of Helsinki. Participants will provide informed consent before enrollment, and all data will be kept confidential and anonymized to protect participants' privacy.

The study findings will be disseminated through peer-reviewed publications, scientific conferences, and presentations to the public, healthcare providers, and patient advocacy groups. The research team aims to leverage the study results to promote awareness, inform clinical practice, and advocate for more equitable access to healthcare and evidence-based interventions for Hispanics/Latinos with MS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Diagnosis of MS
* Relapse-free for at least 30 days
* Able to walk with or without an assistive device
* Insufficient physical activity (i.e., not meeting current physical activity guidelines of 150 minutes of moderate to vigorous physical activity per week)
* Willingness to complete all required testing procedures, outcome questionnaires, and randomization
* Identify as Hispanic/Latino
* Able to speak, read, and understand English
* Currently reside in Chicago
* Access to the internet and email
* Safe for exercise based on the Physical Activity Readiness Questionnaire (PAR-Q)

Exclusion Criteria:

* Not between 18-65 years
* No diagnosis of MS
* Not relapse-free for at least 30 days
* Not able to walk with or without an assistive device
* Too much physical activity (i.e. 150 minutes or more of moderate to vigorous physical activity per week)
* Not willing to complete all required testing procedures, outcome questionnaires, and randomization
* Do not identify as Hispanic/Latino
* Unable to speak, read, and understand English
* Not currently residing in Chicago
* No access to the internet and email
* Not safe for exercise based on the PAR-Q

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-04-27 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Process: Participant Recruitment and Retention | Before, During, and After 16 weeks, pre-, intra- and post-Intervention
  Assessed by recruitment and refusal rates, and retention, attrition, and adherence rates. This will be monitored and assessed with USPS, phone, and electronic mail recruitment, and record all contact with potential participants and refusal reasons. Participants' flow through recruitment, enrollment, and intervention will be monitored, and adherence will be assessed with log books, zoom assessments, and time spent in physical activity as measured during follow-up assessment.
Resources: Communication and Monetary Requirements of the Study | Before, During, and After 16 weeks, pre-, intra- and post-Intervention
  Assessed by communication with participants and staff (needs), and monetary costs of research. This will be monitored and assessed with data collected on initial and follow-up contact with all potential and enrolled participants. A record of all problems and communication alterations will be monitored, as well as all monetary costs for the study that includes both the intervention and control groups.
Management: Data Management and Safety Reporting During the Study | During and After 16 weeks, intra- and post-Intervention
  Assessed by IRB approval procedures, staff preparation and report time for participant communication, time and accuracy in data collection/entry, and reporting and handling of adverse events, serious adverse events, and clinical emergencies. All communications between University IRB and staff, and time from submission of IRB application to approval will be documented. All preparation, call time, attempted call time and report-taking time for each participant during the intervention will be documented. Data completeness, time to record completeness, time to record, enter, and check data will be monitored, and use and handling of all standard university protocol for reporting of all adverse events, serious adverse events, and clinical emergencies will be recorded.
Scientific: Safety, Burden and Treatment Effect of the Study | During and After 16 weeks, intra- and post-Intervention
  Assessed by adverse events, serious adverse events, and clinical emergencies, participants' experience, burden, and compliance during the intervention, and treatment effect. Standard university protocol to record all adverse events, serious adverse events, and clinical emergencies will be followed, and participants will be asked to report all medical concerns for staff to record via log books and zoom chats. Effect size and clinical meaningfulness of any change in physical activity, sedentary behavior, symptoms, and health-related quality of life outcomes will be measured.

SECONDARY OUTCOMES:
Lower Extremity Function | Before and after 16 weeks, baseline and post-intervention
  Assessed by the 30-Second Sit to Stand Test (30STS). The score is the number of complete repetitions of sit-to-stand movements performed for 30 seconds; the minimum value is 0 repetitions, and the maximum value depends on individuals' performance. Higher scores reflect better lower extremity function.
Visual Processing Speed | Before and after 16 weeks, baseline and post-intervention
  Assessed by the Symbol Digit Modalities Test (SDMT). Participants will verbally identify digit-symbol pairings as quickly as possible in response to a series of unpaired symbols displayed on screen. The outcome is the total number of correct responses in 30, 60 and 90 seconds.
Verbal Learning and Memory | Before and after 16 weeks, baseline and post-intervention
  Assessed by the California Verbal Learning Test II (CVLT-II). Participants will be read aloud 16 words and immediately recall as many words as possible, in any order, for each of the five trials. The total score out of 80 will be calculated by summing the number of correct responses from each trial (T1 to T5).
Fatigue Severity | Before and after 16 weeks, baseline and post-intervention
  Assessed by the Fatigue Severity Scale (FSS); scores range between 1 (min) and 7 (max), higher scores reflect greater fatigue severity.
Depressive Symptoms | Before and after 16 weeks, baseline and post-intervention
  Assessed by the Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.
Exercise Behavior | Before and after 16 weeks, baseline and post-intervention
  Assessed by Godin Leisure-Time Exercise Questionnaire (GLTEQ); scores range between 0 (min) and 119 (max), higher scores indicate greater engagement in exercise behavior.
Health-related Quality of Life | Before and after 16 weeks, baseline and post-intervention
  Assessed by the Short Form -12 (SF-12), a shortened version of the short-form 36-item health survey, which measures overall health status.The component scores are adjusted based on a relative average, where a score above 50 is considered above average and a score below 50 is considered below average.

OTHER OUTCOMES:
Social Determinants of Health Factors | Before and after 16 weeks, baseline and post-intervention
  Assessed with the PhenX Toolkit, a consensus measurement for phenotypes and exposures in human research (Cox et al., 2021). Individual SDOH will assess 12 factors (access to health services, health technology, prescription affordability, discrimination in health care, English proficiency, health literacy, job insecurity, neighborhood environment, racial/ethnic discrimination, religious behaviors, spirituality, and wealth), and structural SDOH factors will assess 7 factors (educational attainment, social vulnerability, neighborhood walking and biking environment, water access and sanitation, air quality index, concentrated poverty, and food).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Motl, Ph.D, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flores VA, Silveira SL, Marquez DX, Kinnett-Hopkins D, Miravalle A, Sierra-Morales F, Hernandez-Peraza Z, Motl RW. Rationale for a 4-month, parallel-group, randomized controlled trial to assess the Feasibility and Efficacy of a Remotely delivered exercise training intervention for Hispanics/Latinos with Multiple Sclerosis (FERLA MS). Pilot Feasibility Stud. 2025 May 8;11(1):62. doi: 10.1186/s40814-025-01641-5. PMID 40340698